CLINICAL TRIAL: NCT05270252
Title: Educational Intervention in Nursing Students for the Care of Long-term Cancer Survivors and Their Families: An Exploratory Randomized Controlled Trial
Brief Title: Educational Intervention for Cancer Survivorship Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EICS
Record Dates: First submitted 2022-02-22; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-12

CONDITIONS: Students
Keywords: Long-term survivor, cancer, family; educational intervention, interdisciplinary,; educational methods
MeSH Terms: conditions — Neoplasms | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The study was designed following the framework of the Medical Research Council (MRC) (Craig et al., 2019), for complex interventions.
  The sample size was estimated in at least 58 participants assuming a percentage of potential losses of 10%.
  The recruitment period was from January-February 2021. After receiving permission of the University and approvals from the Ethics Committee (REF. 2020.161), the principal researcher presented the project to the students with a brief oral presentation supported by video. The students who agreed to participate scanned a QR code through which they could request information indicating a contact email.
  Students who requested information, and who met the inclusion criteria, were sent a project information sheet, as well as a Doodle to sign up for the first session. Before the first session, they signed the informed consent and the sociodemographic data were collected through a Google Form questionnaire.
Who Masked: Participant
Masking Description: Participants were blinded in their group assignment; means were put in place to maintain blinding of students throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): no intervention
- Intervention group (Experimental): Interdisciplinary educational intervention with a combination of active educational methods.
  Interventions: Other: Learning and Care

INTERVENTIONS:
Other: Learning and Care — The educational intervention lasted 10 hours: six face-to-face and four for personal study. Three educational methodologies were combined.
  The first: flipped classroom. Students received training material in their email: articles on the needs of families / cancer survivors and family nursing according to the Calgary Model (Wright & Leahey, 2013) and experiential videos of survivors and family members. In the classroom, a week later, a nurse promoted students' self-learning and reflection.
  The second: simulation clinical case. The students received by email a summary of the case and material for their personal work. Students in groups of three performed the entire clinical scenario.
  The third: round table. The components were advanced practice nurse, medical oncologist, cancer survivor and a family member. The content revolved around personal experience in caring for family members and cancer survivors and the interdisciplinary work required for this care.
  Arms: Intervention group

SUMMARY:
The study aims to determine the feasibility and acceptability of an interdisciplinary educational intervention for nursing students to acquire the competence (knowledge, skill and attitude) to care for long-term cancer survivors and their families.

The design is an exploratory randomized controlled trial Following the framework of the Medical Research Council, the method used is a multidisciplinary educational intervention consisting of a flipped classroom, a clinical simulation and a round table with a duration of ten hours. The variables to measure effectiveness were competence and its attributes: knowledge, skills and attitude. The variable to assess acceptability and feasibility was student satisfaction. Data were collected before and after the intervention.

DETAILED DESCRIPTION:
The study was designed following the framework of the Medical Research Council (MRC) , for complex interventions. The study participants were 3rd-year Nursing bachelor students from the University of Navarra (Spain). The educational intervention was called Learning & Care, and it was framed within the European Higher Education Area.

For the design of the intervention, the following steps were followed within the MRC framework: (1) review of the literature to know the educational methodologies used in the field of health for the care of patients with cancer and exploration of the different conceptual models of family nursing, (2) design and development of an educational intervention proposal developed by the researchers of the study, and (3) the evaluation of the intervention proposal by a multidisciplinary Expert Panel composed of 11 members: five nurses (primary care, researchers, teachers and hospitalization), a medical oncologist, a psycho-oncologist, a pharmacist, a student, a cancer survivor and a family member of a cancer survivor. With the suggestions of the panel, the final educational intervention was developed, and the exploratory and piloting study was carried out.

The data collection lasted from February to April 2021, a period in which the students did not have exams. Sociodemographic information of all participants (intervention and control group) was collected only at baseline using a researcher-developed questionnaire that included variables such as: age, sex, previous study of some degree (it is common in Spain to do double degrees), previous courses or training related to family nursing and experience as healthcare worker (this last information was collected because some students work as nursing assistants while studying the Bachelor's degree).

In addition, data was collected on the level of knowledge, skills and attitude of the students to carry out care focused on the cancer survivor and his family, both in the Control group (CG) and in the Intervention group (IG) before and after the educational intervention with the IG. At the end of the training with the IG, the data from the IG and GC on student satisfaction were collected.

The students completed the sociodemographic information and the data on knowledge and attitude through the online platform Google Form. The principal researcher collected the data on the students' skills on a tablet. Lastly, the level of student satisfaction with the program was collected on site and on paper once the training program was completed.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the 3rd year of nursing at the Faculty of Nursing of the University of Navarra and who voluntarily agree to participate in the study

Exclusion Criteria:

* 1st and 2nd year nursing students since they had not had contact with clinical practice.
* 4th year nursing students due to being in a clinical practice period and being outside the institution where the intervention was carried out.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Knowledge | February-April (3 months)
  To assess the level of knowledge acquired by students about the needs of long-term survivors and their families, as well as about family nursing and family assessment and intervention tools according to the Calgary Model, an ad hoc multiple choice test was designed. 20 multiple choice questions. The test was piloted among team members and students to validate their understanding and identify possible errors in multiple responses.
Skills | February-April (3 months)
  The Van Gelderen Family-Care Rubric Scale (VGFCR) was used (Van Gelderen et al., 2019). The VGFCR is made up of 12 evaluable items, each one between 1 and 3 points. The scale groups the items into two groups: communication in the family and the family as a client. In each of the groups you can get a maximum score of 18 points. The total skill value is 36. In general, reliable VGFCR was determined with Fleiss' Kappa significance at p = 0.05 at the 95% confidence interval and Cronbach's alpha 0.842. This scale is available in English, permission was requested from the author to translate it into Spanish and I use the study. The linguistic-cultural adaptation was carried out through the direct and inverse translation methodology (Bracken & Barona, 1991). Once the double translation was done, the scale translated into Spanish was sent to the main author, who agreed.
Attitude | February-April (3 months)
  To measure attitude, the FINC-NA scale (Barreto et al., 2022) was used, which has been widely used to measure the attitude of nurses to involve families in care. The scale consists of 26 evaluable items in a range between 1 and 4 points, organized into 4 groups: (1) Family as another resource for nursing care, (2) Family as collaborator in dialogue, (3) Family as burden and ( 4) Family as their own resource. For the calculation of the "family as a burden" group, the data were inverted (Hagedoorn et al., 2020). The total value of the attitude scale is 104 points. This scale is validated in Spanish in a sample of 274 professionals and obtained a total Cronbach's alpha coefficient of 0.864 for the total scale, ranging between 0.888 and 0.769 in the subscales. The factorial analysis identified 4 factors that explained 54.22% of the total variance (Pascual Fernandez et al., 2015).

SECONDARY OUTCOMES:
student satisfaction | February-April (3 months)
  For the evaluation of the secondary variable, student satisfaction with the Learning & Care intervention, the Client Satisfaction Questionnaire (CSQ-8) (Echeburua & Corral, 2010) was used. This questionnaire consists of 8 items and has been validated in Spanish with very high levels of internal consistency, according to Cronbach's coefficients, which range between 0.83 and 0.93.(Echeburua & Corral, 2010; Martinez-Azurmenti & Beitia Fernandez, 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Marta Domingo, Principal Investigator — Clinica Universidad de Navarra, Universidad de Navarra
Locations (1):
- Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Wright LM. Brain science and illness beliefs: an unexpected explanation of the healing power of therapeutic conversations and the family interventions that matter. J Fam Nurs. 2015 May;21(2):186-205. doi: 10.1177/1074840715575822. Epub 2015 Mar 12. PMID 25766206
- [Background] Gelderen, S. Van, Engebretson, A., Miller, A., Hancock, A., Ehmke, S., Swan, M., & Garrow, A. (2019). A Family-Care Rubric : Developing Family Care and Communication Skills Using Simulation. Clinical Simulation in Nursing, 36, 47-58. https://doi.org/10.1016/j.ecns.2019.07.006
- [Background] Bracken, B. A., & Barona, A. (1991). State of the Art Procedures for Translating, Validating and Using Psychoeducational Tests in Cross-Cultural Assessment. School Psychology International, 12(April 1991), 119-132. https://doi.org/10.1177/0143034391121010
- [Background] Barreto MDS, Marquete VF, Camparoto CW, Garcia-Vivar C, Barbieri-Figueiredo MDC, Marcon SS. Factors associated with nurses' positive attitudes towards families' involvement in nursing care: A scoping review. J Clin Nurs. 2022 Dec;31(23-24):3338-3349. doi: 10.1111/jocn.16226. Epub 2022 Jan 26. PMID 35083808
- [Background] Hagedoorn EI, Paans W, Jaarsma T, Keers JC, van der Schans CP, Luttik MLA. The importance of families in nursing care: attitudes of nurses in the Netherlands. Scand J Caring Sci. 2021 Dec;35(4):1207-1215. doi: 10.1111/scs.12939. Epub 2020 Dec 3. PMID 33270268
- [Result] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Result] Domingo-Osle M, La Rosa-Salas V, Ambrosio L, Elizondo-Rodriguez N, Garcia-Vivar C. Educational methods used in cancer training for health sciences students: An integrative review. Nurse Educ Today. 2021 Feb;97:104704. doi: 10.1016/j.nedt.2020.104704. Epub 2020 Dec 7. PMID 33352353
- [Derived] Domingo-Osle M, La Rosa-Salas V, Garcia-Vivar C. Educational Intervention for Family Nursing Students in Long-Term Cancer Survivorship: A Randomized Pilot Trial. J Fam Nurs. 2023 Aug;29(3):248-262. doi: 10.1177/10748407231167438. Epub 2023 May 21. PMID 37211798